CLINICAL TRIAL: NCT06246513
Title: A Phase 3 Multinational, Open-label, Systemic Gene Delivery Study to Evaluate the Safety and Efficacy of SRP-9003 in Subjects With Limb Girdle Muscular Dystrophy 2E/R4
Brief Title: A Trial to Learn More About an Experimental Gene Therapy Called Bidridistrogene Xeboparvovec (SRP-9003) as a Possible Treatment for Limb Girdle Muscular Dystrophy 2E/R4
Acronym: EMERGENE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9003-301; 2022-503112-17-00 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Limb-girdle Muscular Dystrophy
Keywords: Limb Girdle Muscular Dystrophy Type 2E/R4; LGMD2E/R4; Pediatric; SRP-9003; scAAVrh74.MHCK7.hSGCB; bidridistrogene xeboparvovec; Non-ambulatory; Ambulatory
MeSH Terms: conditions — Muscular Dystrophies, Limb-Girdle | interventions — Glucocorticoids; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRP-9003 (Experimental): Participants will receive a single intravenous (IV) infusion of SRP-9003.
  Interventions: Biological: SRP-9003; Drug: Glucocorticoid

INTERVENTIONS:
Biological: SRP-9003 — Solution for single IV infusion
  Other Names: scAAVrh74.MHCK7.hSGCB, bidridistrogene xeboparvovec
Drug: Glucocorticoid — Oral tablet (prophylactic)
  Other Names: Prednisone or equivalent

SUMMARY:
This is a multicenter, global study of the effects of a single systemic dose of SRP-9003 on beta-sarcoglycan (β-SG) gene expression in participants with limb-girdle muscular dystrophy, type 2E/R4 (LGMD2E/R4). This study will consist of both ambulatory participants (Cohort 1) and non-ambulatory participants (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1, only ambulatory participants:

  * Able to walk without assistive aid
  * 10-meter walk test (10MWT) <30 seconds
  * NSAD ≥25
* Cohort 2, only non-ambulatory participants:

  * 10MWT ≥30 seconds or unable to perform
  * PUL 2.0 entry scale score ≥3
* Participants must possess 1 homozygous or 2 heterozygous pathogenic and/or likely pathogenic β-SG DNA gene mutations
* Able to cooperate with muscle testing
* Participants must have adeno-associated virus serotype rh74 (AAVrh74) antibody titers <1:400 (that is, not elevated) as determined by AAVrh74 antibody enzyme-linked immunosorbent assay.

Exclusion Criteria:

* Left ventricular ejection fraction < 40% or clinical signs and/or symptoms of cardiomyopathy
* Forced vital capacity ≤40% of predicted value and/or requirement for nocturnal ventilation
* Diagnosis of (or ongoing treatment for) an autoimmune disease and on active immunosuppressant treatment
* Presence of any other clinically significant illness or medical condition (other than LGMD2E/R4)

Other inclusion/exclusion criteria apply.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-03-04 (Actual); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Change from Baseline in β-SG Expression at Day 60 Post-dose as Measured by Immunofluorescence (IF) Percent β-SG Positive Fibers | Baseline, Day 60

SECONDARY OUTCOMES:
Cohort 1 and Cohort 2: Change From Baseline in β-SG Expression at Day 60 Post-dose as Measured by Western Blot | Baseline, Day 60
Cohort 1 and Cohort 2: Change From Baseline in β-SG Expression at Day 60 Post-dose as Measured by IF Percent Fluorescent Intensity (PFI) | Baseline, Day 60
Cohort 2: Change From Baseline in β-SG Expression at Day 60 Post-dose as Measured by IF Percent β-SG Positive Fibers (PβSGPF) | Baseline, Day 60
Cohort 1 and Cohort 2: Change From Baseline Through Month 60 in North Star Assessment for Dysferlinopathy (NSAD) Total Score | Baseline through Month 60
Cohort 1 and Cohort 2: Change From Baseline Through Month 60 in Performance of Upper Limb Version 2.0 (PUL 2.0) Total Score | Baseline through Month 60
Cohort 1: Change From Baseline Through Month 60 in the Time to Rise from the Floor Test | Baseline through Month 60
Cohort 1: Change From Baseline Through Month 60 in the Time to Complete the 10-meter Walk/Run (10MWR) Test | Baseline through Month 60
Cohort 1: Change From Baseline Through Month 60 in the Time to Ascend 4 Steps Test | Baseline through Month 60
Cohort 1: Change From Baseline Through Month 60 in the Time to Complete the 100-meter Walk/Run (100MWR) Test | Baseline through Month 60
Cohort 1: Change From Baseline Through Month 60 in the Timed Up and Go Test | Baseline through Month 60
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Baseline through Month 60
Change From Baseline Through Month 60 in Creatine Kinase Level | Baseline through Month 60
Time to Change of Loss of Ambulation | Baseline through Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (10):
- United States (4):
  - University of California, San Diego-Altman Clinical and Translational Research Institute, La Jolla, California
  - Nationwide Childrens Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of The King's Daughter, Norfolk, Virginia
- Belgium (2):
  - University Hospital Leuven (UZ Leuven), Leuven, Vlaams Brabant
  - NMRC Gent (UZ Gent), Ghent
- Universitatsklinikum Essen; Kinderklinik I, Sozialpadiatrisches Zentrum, Essen, North Rhine-Westphalia, Germany
- Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan, Italy
- Hospital Sant Joan de Deu, Barcelona, Spain
- Newcastle University, Newcastle upon Tyne, United Kingdom